CLINICAL TRIAL: NCT00795340
Title: A Double Blind Randomized Trial of Cediranib Versus Placebo in Patients Receiving Paclitaxel/Carboplatin Chemotherapy for the Treatment of Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Cediranib, Paclitaxel, and Carboplatin in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR29; CAN-NCIC-BR29; CDR0000618671 (Other: PDQ)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2015-06

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; cediranib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I Cediranib (Experimental): Patients receive oral cediranib once daily on days 1-21 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.
  Interventions: Drug: carboplatin; Drug: cediranib maleate; Drug: paclitaxel
- Arm II Placebo (Placebo Comparator): Patients receive oral placebo once daily on days 1-21 and paclitaxel and carboplatin as in arm I.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Other: placebo

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: cediranib maleate — Given orally
  Arms: Arm I Cediranib
Drug: paclitaxel — Given IV
Other: placebo — Given orally
  Arms: Arm II Placebo

SUMMARY:
RATIONALE: Cediranib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether cediranib is more effective than a placebo when given together with paclitaxel and carboplatin in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying how well cediranib works when given together with paclitaxel and carboplatin in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare overall survival of patients with stage IIIB-IV non-small cell lung cancer treated with cediranib vs placebo administered in combination with paclitaxel and carboplatin.

Secondary

* To compare the progression-free survival of patients treated with these regimens.
* To compare the objective response rates in patients treated with these regimens.
* To estimate time to response and response duration in patients treated with these regimens.
* To evaluate the nature, severity, and frequency of toxicities, including hemorrhage and hemoptysis, in patients treated with these regimens.
* To compare the pharmacokinetics of paclitaxel between the two arms in a subset of enrolled patients
* To compare the quality of life of patients treated with these regimens.
* To determine the incremental cost effectiveness and cost utility ratios for these regimens.
* To correlate the expression of tissue markers (at diagnosis) with outcomes and response in an exploratory fashion OUTLINE: This is a multicenter study. Patients are stratified by gender, center, disease stage (IIIB vs IV), weight loss (< 5% vs 5-10% vs unknown), and prior adjuvant chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.
* Arm I: Patients receive oral cediranib once daily on days 1-21 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.
* Arm II: Patients receive oral placebo once daily on days 1-21 and paclitaxel and carboplatin as in arm I.

Treatment in both arms repeats every 21 days for 4 to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on day 1 of each course, and periodically thereafter.

After completion of study therapy, patients are followed every 12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically* confirmed non-small cell carcinoma of the lung

  * Stage IIIB or IV disease NOTE: *Diagnosis by sputum cytology alone allowed provided it is confirmed by a second sputum specimen
* Measurable disease, defined as at least 1 measurable lesion > 20 mm by x-ray, ultrasound, or physical exam or ≥ 10 mm (lymph nodes must be ≥ 15 mm in the short axis) by spiral CT scan or physical exam (in the first 260 patients randomized**)

  * Measurable lesions that are sole sites of disease must be outside a previous radiotherapy field unless disease progression has been documented NOTE: **Measurable or nonmeasurable disease allowed after the first 260 patients
* No appreciable cavitation in central thoracic lesions
* No untreated brain or meningeal metastases

  * Patients with treated and radiologic or clinical evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible provided the metastases are asymptomatic and do not require corticosteroids
* No pleural effusion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance > 50 mL/min
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2 times ULN (< 5 times ULN if due to liver metastasis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception (barrier method for men)
* No other malignancy within the past 5 years, except in situ cancer, basal cell or squamous cell skin cancer, or malignancy cured by definitive prior therapy alone (e.g., surgery) and continuously disease-free for at least 5 years
* Mean QTc with Bazett correction ≤ 480 msec in screening ECG (at least one value must be ≤ 480 msec when measured automatically or manually corrected using Bazett's or Fridericia's correction)
* No history of familial long QT syndrome
* No untreated and/or uncontrolled cardiovascular conditions and/or symptomatic cardiac dysfunction including any of the following:

  * Unstable angina
  * Congestive heart failure
  * Myocardial infarction within the past year
  * Cardiac ventricular arrhythmias requiring medication
  * History of second or third degree atrioventricular conduction defects
* LVEF > 50% in patients with significant cardiac history, even if controlled
* No resting BP consistently > 150 mm Hg systolic and/or > 100 mm Hg diastolic
* No poorly controlled hypertension
* No history of labile hypertension or poor compliance with anti-hypertensive medication
* No overt bleeding (> 30 mL bleeding/episode) from any site within the past 3 months
* No clinically relevant hemoptysis (> 5 mL fresh blood) within the past 4 weeks

  * Flecks of blood in sputum allowed
* No active or uncontrolled infections, or serious illnesses or medical conditions which would not permit the patient to be treated according to the study
* No prior allergic reactions to drugs containing Cremophor EL®
* No inflammatory bowel disease (e.g., Crohn disease or ulcerative colitis)
* No documented weight loss > 10% within the past 3 months

  * Patients with weight loss 5-10% or whose weight loss status is unknown are eligible provided serum albumin levels are ≥ 30 g/L
* No peripheral neuropathy > grade 1
* Must be fit for combined modality treatment
* Sufficiently fluent and willing to complete quality-of-life questionnaires

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* No prior chemotherapy for metastatic or recurrent disease
* No prior anti-angiogenic therapy (e.g., bevacizumab, cediranib, AZD6474, PTK/ZK, sunitinib malate, or other agents considered angiogenesis inhibitors by NCIC Clinical Trials Group for any indication)

  * Prior cox-2 inhibitors in standard doses allowed
* At least 12 months since prior adjuvant chemotherapy for completely resected disease

  * Combined chemotherapy/radiotherapy regimens for locally advanced stage IIIB disease not allowed
* At least 21 days since prior radiotherapy
* At least 21 days since prior cetuximab or other monoclonal antibodies
* At least 14 days since prior EGFR inhibitor therapy for adjuvant therapy or metastatic disease (e.g., tyrosine kinase inhibitors, vaccines, or other agents considered by NCIC CTG as acting on the EGFR pathway)
* At least 14 days since prior major surgery
* At least 1 week since prior corticosteroids
* No other concurrent experimental drugs, anticancer treatment, or investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-02-04 (Actual); Primary Completion 2012-01-09 (Actual); Study Completion 2014-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. Laurie, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (19):
- Brazil (2):
  - Instituto Nacional de Cancer (INCA), Rio de Janeiro
  - Instituto de Cancer Arnaldo Vieira de Carvalho, São Paulo
- Canada (17):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec
  - University Institute of Cardiology and, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laurie SA, Solomon BJ, Seymour L, Ellis PM, Goss GD, Shepherd FA, Boyer MJ, Arnold AM, Clingan P, Laberge F, Fenton D, Hirsh V, Zukin M, Stockler MR, Lee CW, Chen EX, Montenegro A, Ding K, Bradbury PA. Randomised, double-blind trial of carboplatin and paclitaxel with daily oral cediranib or placebo in patients with advanced non-small cell lung cancer: NCIC Clinical Trials Group study BR29. Eur J Cancer. 2014 Mar;50(4):706-12. doi: 10.1016/j.ejca.2013.11.032. Epub 2013 Dec 17. PMID 24360368

RESULTS

PARTICIPANT FLOW:
Groups:
- Cediranib: Patients receive oral cediranib once daily on days 1-21 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.
  carboplatin: Given IV
  cediranib maleate: Given orally
  paclitaxel: Given IV
- Placebo: Patients receive oral placebo once daily on days 1-21 and paclitaxel and carboplatin as in arm I.
  carboplatin: Given IV
  paclitaxel: Given IV
  placebo: Given orally
Period: Overall Study
Arm/Group | Cediranib | Placebo
Started | 153 | 153
Completed | 146 | 153
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib | Placebo | Total
Number analyzed (Participants) | 153 | 153 | 306
Age, Continuous [Median (Full Range); unit: years] | 63 [23 to 85] | 62 [36 to 77] | 62 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 84 | 83 | 167
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 129 | 132 | 261
  Hispanic | 1 | 2 | 3
  Black | 1 | 5 | 6
  Asian | 12 | 9 | 21
  Aboriginal | 1 | 0 | 1
  Other | 7 | 2 | 9
  Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 102 | 98 | 200
  Brazil | 7 | 11 | 18
  Australia | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Medians of survival time, and their confidence intervals.
Time Frame: at every 3 months visit throughout trial, a median of 13.1 months.
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cediranib | Placebo
Number analyzed (Participants) | 153 | 153
months | 12.2 [9.1 to 18.0] | 12.1 [11.1 to 15.5]

2. Secondary Outcome: Progression-free Survival
Description: Medians of PFS and their confidence intervals by arm
Time Frame: at every 3 months visit throughout trial, a median of 12 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cediranib | Placebo
Number analyzed (Participants) | 153 | 153
months | 5.52 [4.86 to 6.05] | 5.45 [4.86 to 5.78]

3. Secondary Outcome: Objective Tumor Response as Assessed by RECIST Criteria v1.1.
Description: Every 6 weeks at the end of every 2 cycles during protocol treatment and every 12 weeks after protocol treatment until progression.
Time Frame: Every 6 weeks at the end of every 2 cycles during protocol treatment and every 12 weeks after protocol treatment until progression.
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cediranib | Placebo
Number analyzed (Participants) | 153 | 153
percentage of participants | 52 [44 to 60] | 34 [26 to 42]

ADVERSE EVENTS:
Time Frame: from the start of treatment to time of 4 weeks after stopped the treatment.
Groups:
- Cediranib: Patients receive oral cediranib once daily on days 1-21 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.
- Placebo: Patients receive oral placebo once daily on days 1-21 and paclitaxel and carboplatin as in arm I.
Arm/Group | Cediranib | Placebo
Serious Adverse Events (participants affected / at risk) | 67/153 | 54/153
Other Adverse Events (participants affected / at risk) | 151/153 | 152/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib (N=153) | Placebo (N=153)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 7
Hemoglobin (Blood and lymphatic system disorders) | 1 | 3
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 1
Cardiopulmonary arrest (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular arrhythmia Atrial fibrillation (Cardiac disorders) | 0 | 1
Supraventricular arrhythmia Sinus tachycardia (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Blurred vision (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 0
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 5
Obstruction, GI Small bowel NOS (Gastrointestinal disorders) | 1 | 0
Pain Abdomen NOS (Gastrointestinal disorders) | 3 | 0
Perforation, GI Colon (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 5
Death Death NOS (General disorders) | 1 | 2
Death Disease progression NOS (General disorders) | 6 | 4
Edema: limb (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Fever (General disorders) | 0 | 5
Pain Chest/thorax NOS (General disorders) | 1 | 4
Pain Liver (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 3
Colitis, infectious (Infections and infestations) | 1 | 0
Infection (documented clinically) Blood (Infections and infestations) | 1 | 0
Infection (documented clinically) Colon (Infections and infestations) | 0 | 1
Infection (documented clinically) Lung (Infections and infestations) | 2 | 2
Infection (documented clinically) Meninges (Infections and infestations) | 1 | 0
Infection (documented clinically) Skin (Infections and infestations) | 0 | 1
Infection (documented clinically) Upper airway NOS (Infections and infestations) | 4 | 0
Infection with normal ANC Abdomen NOS (Infections and infestations) | 2 | 0
Infection with normal ANC Anal/perianal (Infections and infestations) | 1 | 0
Infection with normal ANC Bladder (Infections and infestations) | 2 | 0
Infection with normal ANC Colon (Infections and infestations) | 1 | 1
Infection with normal ANC Larynx (Infections and infestations) | 1 | 0
Infection with normal ANC Lung (Infections and infestations) | 5 | 7
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Thrombosis/embolism (vascular access) (Injury, poisoning and procedural complications) | 0 | 2
Neutrophils (Investigations) | 0 | 4
Platelets (Investigations) | 1 | 1
cTnI (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Muscle weakness Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain Back (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain Bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain Muscle (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CNS hemorrhage (Nervous system disorders) | 1 | 0
CNS ischemia (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 2
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Neuropathy: cranial CN VIII (Nervous system disorders) | 0 | 1
Pain Head/headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 3 | 1
Hemorrhage, GU Urinary NOS (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hemorrhage pulmonary Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage - Other (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 11 | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib (N=153) | Placebo (N=153)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 8
Supraventricular arrhythmia Sinus tachycardia (Cardiac disorders) | 1 | 8
Hearing (without monitoring program) (Ear and labyrinth disorders) | 4 | 8
Blurred vision (Eye disorders) | 15 | 11
Constipation (Gastrointestinal disorders) | 87 | 101
Diarrhea (Gastrointestinal disorders) | 120 | 56
Dry mouth (Gastrointestinal disorders) | 7 | 11
Dysphagia (Gastrointestinal disorders) | 8 | 4
Heartburn (Gastrointestinal disorders) | 28 | 31
Hemorrhoids (Gastrointestinal disorders) | 9 | 3
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 25 | 15
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 36 | 21
Nausea (Gastrointestinal disorders) | 102 | 95
Pain Abdomen NOS (Gastrointestinal disorders) | 34 | 27
Vomiting (Gastrointestinal disorders) | 56 | 59
Edema: limb (General disorders) | 21 | 25
Fatigue (General disorders) | 127 | 120
Fever (General disorders) | 9 | 22
Flu-like syndrome (General disorders) | 11 | 7
Pain Chest/thorax NOS (General disorders) | 38 | 43
Allergic reaction (Immune system disorders) | 13 | 23
Infection with normal ANC Lung (Infections and infestations) | 12 | 8
Infection with normal ANC Upper airway NOS (Infections and infestations) | 15 | 15
Infection with normal ANC Urinary tract NOS (Infections and infestations) | 8 | 11
Infection with unknown ANC Upper airway NOS (Infections and infestations) | 10 | 5
Bruising (Injury, poisoning and procedural complications) | 8 | 5
Weight loss (Investigations) | 35 | 11
Anorexia (Metabolism and nutrition disorders) | 93 | 77
Dehydration (Metabolism and nutrition disorders) | 14 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 8
Muscle weakness Extremity-lower (Musculoskeletal and connective tissue disorders) | 14 | 9
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 7 | 10
Pain Back (Musculoskeletal and connective tissue disorders) | 40 | 38
Pain Bone (Musculoskeletal and connective tissue disorders) | 27 | 27
Pain Chest wall (Musculoskeletal and connective tissue disorders) | 17 | 20
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 34 | 24
Pain Joint (Musculoskeletal and connective tissue disorders) | 58 | 67
Pain Muscle (Musculoskeletal and connective tissue disorders) | 55 | 75
Pain Neck (Musculoskeletal and connective tissue disorders) | 8 | 8
Pain Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 19
Dizziness (Nervous system disorders) | 37 | 29
Memory impairment (Nervous system disorders) | 10 | 4
Neuropathy-motor (Nervous system disorders) | 15 | 9
Neuropathy-sensory (Nervous system disorders) | 110 | 110
Pain Head/headache (Nervous system disorders) | 49 | 35
Taste alteration (Nervous system disorders) | 32 | 26
Confusion (Psychiatric disorders) | 7 | 10
Insomnia (Psychiatric disorders) | 46 | 53
Mood alteration Anxiety (Psychiatric disorders) | 27 | 33
Mood alteration Depression (Psychiatric disorders) | 13 | 21
Urinary frequency (Renal and urinary disorders) | 9 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 107 | 108
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 104 | 92
Hemorrhage pulmonary Lung (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Hemorrhage pulmonary Nose (Respiratory, thoracic and mediastinal disorders) | 35 | 12
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pain Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Voice changes (Respiratory, thoracic and mediastinal disorders) | 29 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 121 | 116
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 11
Hand-foot (Skin and subcutaneous tissue disorders) | 11 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 15
Rash (Skin and subcutaneous tissue disorders) | 47 | 36
Sweating (Skin and subcutaneous tissue disorders) | 6 | 10
Hypertension (Vascular disorders) | 77 | 21
Hypotension (Vascular disorders) | 8 | 7
Thrombosis/thrombus/embolism (Vascular disorders) | 16 | 15

LIMITATIONS AND CAVEATS:
Early termination at phase II part of the trial, leading to small numbers of subjects analyzed, and limited follow up time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes